CLINICAL TRIAL: NCT04905888
Title: Hyperbaric Oxygen Therapy for Long COVID Patients With Pulmonary Sequela - Pilot Study
Brief Title: Hyperbaric Oxygen for Long COVID-19 Pulmonary Sequela
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Closure/ move of MRI facility.
Sponsor: Peter Lindholm (Other)
Responsible Party: Sponsor-Investigator, Peter Lindholm, Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRPP210260
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Covid19
Keywords: hyperbaric oxygen; hyperbaric oxygen therapy; long covid
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: hbo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Hyperbaric oxygen therapy (Experimental): Treatment with hyperbaric oxygen
  Interventions: Combination Product: Hyperbaric oxygen therapy
- Control (No Intervention): Control, no treatment.

INTERVENTIONS:
Combination Product: Hyperbaric oxygen therapy — Subjects randomized to treatment will receive up to ten 90 minute treatments with hyperbaric oxygen over a 2-3 week period.
  Arms: Hyperbaric oxygen therapy

SUMMARY:
This is a pilot study in 24 subjects where half will be randomized to 10 treatments with hyperbaric oxygen (HBO). It will primarily study pulmonary sequelae with imaging and physiological measurements (low dose chest computer tomography (CT), Ventilation/perfusion with magnetic resonance imaging (VA/Q MRI), cardiopulmonary exercise testing with pulse oximetry (SpO2) and spirometry including diffusion capacity for carbon monoxide (DLCO). The target patient group will be previously healthy whom have had covid-19 with lingering symptoms past 12 weeks of recovery from the acute phase.

DETAILED DESCRIPTION:
Long COVID or Post-Acute Sequelae of SARS-CoV-2 infection (PASC) is current terms for patients demonstrating fatigue, chest pain, exertion malaise, dyspnea, cognitive dysfunction, and headaches, just to name a few symptoms that can last more than 12-weeks after the initial infection of SARS-CoV-2. Pulmonary symptoms of dyspnea and exercise intolerance may be due to pulmonary gas exchange derangement, which could be from hypoxic pulmonary vasoconstriction (HPV) inhibition due to lingering inflammatory processes. Hyperbaric oxygen (HBO) has known anti-inflammatory effects, shown in multiple organ systems, and recently reported in case studies to improve outcomes of acute COVID-19 pneumonitis. If there is pulmonary inflammation it is possible that HBO can improve pulmonary gas exchange by restoring HPV. To test this hypothesis, we plan to perform a mechanistic study on V̇A/Q̇ matching in Long COVID patients with lingering pulmonary symptoms. The etiology of symptoms is unknown, but it is probable that the inflammatory processes associated with COVID-19 may inhibit HPV.

This is an open, randomized, controlled clinical trial with hyperbaric oxygen therapy delivered by a hyperbaric chamber as the intervention. Twelve patients will receive ten HBO therapy (HBOT) over a 2-3-week period, and twelve patients will serve as controls and receive no HBOT. Each HBOT session will administer oxygen (O2) at 2.4 atmospheres absolute pressure (ATA) (100% O2) for 90 minutes in a hyperbaric chamber.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years old
* COVID-19 at least 12 weeks prior, +PCR test and/or documented clinical symptoms
* Desaturate to <94% during the 6-MWT and/or have abnormal spirometry or DLCO values below the lower limit of normal (LLN)
* Active life-style before contracting COVID-19

Exclusion Criteria:

* Pregnant or lactating women
* Individuals that are unable walk or get in and out of bed by themselves
* Weighing over 300 lbs. or Body mass index (BMI) >30
* Inability to provide written informed consent
* Inability or unwillingness to adhere to 10 HBOT treatment sessions over a 2 to 3 week- time period or to complete follow up questionnaires/telephone contacts.
* Claustrophobia and inability to enter the hyperbaric chamber for session.
* Inability to effectively equalize the middle ear during ambient pressure changes. History of tympanic membrane perforation, head and neck surgery with compromised Eustachian tube function, including tracheostomy, mastoidectomy, middle ear surgical procedures and cochlear implants.
* History of pulmonary disease prior to COVID-19 including asthma, chronic obstructive pulmonary disease (COPD), bullous lung disease, previous thoracotomy, pneumothorax or history of pneumothorax prior to having COVID-19.
* History of cardiovascular disease prior to having COVID-19.
* History of type 1 or 2 diabetes prior to having COVID-19
* History of neurovascular diseases (e.g. recent stroke) prior to having COVID-19
* History of uncontrolled hypertension prior to having COVID-19
* History of retinitis pigmentosa prior to having COVID-19
* History of renal disease prior to having COVID-19
* History of seizure disorder prior to having COVID-19
* Active or uncontrolled cancer diagnosis.
* Active or uncontrolled psychiatric disease.
* Acute upper respiratory tract infection
* History of exposure to bleomycin
* Taking the following concomitant medications: PDE5 inhibitors, carbonic anhydrase inhibitors, beta blockers, alpha blockers, nitrates.
* MRI incompatibilities- a cardiac pacemaker, metal fragments in the eyes, skin, body; heart valve replacement, brain clips, venous umbrella, intercranial bypass, renal, aortic clips, prosthetic devices for middle ear, eye, joint or penile implants, joint replacements; hearing aid, neurostimulator, insulin pump, I.U.D, pregnant or trying to become pregnant, shunts/stents, metal mesh/coil implants; metal plate/pin/screws/wires, any other implants; permanent eyeliner/eyebrows with metal containing dyes, dental work within 6 weeks, claustrophobia.
* Involved in another clinical trial that does not allow enrollment in other clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Exercise tolerance | 3 months
  Cardiopulmonary exercise testing with pulse oximetry and maximal oxygen uptake,VO2max (ml/kg/min)

SECONDARY OUTCOMES:
Excercise tolerance walk test | 3 months
  6 minute walk test, in meters
Dyspnea perception 1 | 3 Months
  UCSD Shortness of breath (SOB) 24 questions using a 0-6-point scale per question Total score (0-120) The higher the score the greater the dyspnea
Dyspnea perception 2 | 3 Months
  PROMIS dyspnea questionnaire/scales (Patient-Reported Outcomes Measurement Information System).
  Shortness of Breath in general (0-10) Intensity of Shortness of breath (0-10) Frequency of Shortness of breath (0-10) Duration of Shortness of breath (0-10) The higher the score the greater the dyspnea
Pulmonary function test 1 | 3 months
  Spirometry FEV1 (L) FEV1 %predicted FVC (L) FVC %predicted PEF (l/Min) PEF %predicted
Pulmonary function test 2 | 3 months
  Lung Diffusion Capacity DLCO (ml/min/mmHg) DLCO %predicted
V̇A/Q̇ matching measured with magnetic resonance imaging | 3 months
  pulmonary ventilation/perfusion matching with Lung heterogeneity expressed as relative dispersion in ventilation and perfusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No